CLINICAL TRIAL: NCT03192163
Title: Cultural, Racial, and Ethnic Differences in Treatment Preferences and Perceptions of Acne Vulgaris
Brief Title: Cultural Differences in Treatment Preferences and Perceptions of Acne
Acronym: CDTPPA
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: STU00205213
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ResearchMatch Group
  Interventions: Other: Survey
- Northwestern Center for Ethnic Skin Group
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — 31 question survey with questions regarding non-identifying demographic information such as age and gender. This survey also contains questions about acne treatment preferences, racial/ethnic background, and cultural identity in addition to a few Willingness to Pay questions.

SUMMARY:
This study will use a survey to examine relationships between culture, race, and ethnicity with treatment preferences and perceptions for acne vulgaris.

DETAILED DESCRIPTION:
The purpose of this study is to determine how explanatory models, perceptions, and treatment preferences of acne vulgaris vary across different cultures and racial and ethnic backgrounds. This study will also use Willingness to Pay to investigate differences in treatment valuation. Clarifying these differences will better inform patient counseling and treatment adherence by improving the quality of shared decision making.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have acne vulgaris, be at least 18 years of age, and must be able to complete a survey published in English.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Acne vulgaris in the US
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Willingness to Pay | 15 minutes
  percentage of income individual is willing to pay to use a treatment that improves his or her acne
Preferred and Least Preferred Treatments | 15 minutes
  ranked list of treatments for acne that individuals prefer and don't prefer using (ie. masks/facials, isotretinoin, etc) and reasons for why individuals prefer or don't prefer using that treatment (ie. cost, safety, efficacy, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Survey — http://j.mp/2qdz7P2 — This is the RedCap survey that subjects will take.